CLINICAL TRIAL: NCT00126464
Title: A Pilot Clinical Trial to Evaluate the Biological Activity of Fulvestrant (Faslodex) in Breast Ductal Carcinoma (DCIS)
Brief Title: Fulvestrant or Tamoxifen in Treating Postmenopausal Women Who Are Undergoing Surgery for Ductal Carcinoma in Situ of the Breast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000430705; CSMC-00000244; CSMC-4415/CR00000244; ZENECA-CSMC-00000244; CSMC-1B-03-7
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2006-07

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Fulvestrant; Tamoxifen; Neoadjuvant Therapy

INTERVENTIONS:
Drug: fulvestrant
Drug: tamoxifen citrate
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant or tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving fulvestrant or tamoxifen before surgery may be an effective treatment for breast cancer.

PURPOSE: This randomized clinical trial is studying how well giving fulvestrant or tamoxifen works in treating postmenopausal women who are undergoing surgery for ductal carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine, preliminarily, the efficacy of neoadjuvant fulvestrant, in terms of molecular changes in markers of the estrogen pathway, cell proliferation and apoptosis, and the epidermal growth factor pathway, in postmenopausal women with newly diagnosed ductal carcinoma in situ of the breast.

Secondary

* Determine the toxicity profile of fulvestrant in these patients.

OUTLINE: This is a randomized, placebo-controlled, pilot, multicenter study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral placebo once daily on days 1-21.
* Arm II: Patients receive oral tamoxifen once daily on days 1-21.
* Arm III: Patients receive fulvestrant intramuscularly (IM) on day 1.
* Arm IV: Patients receive fulvestrant IM as in arm III but at a higher dose. In all arms, treatment continues in the absence of disease progression or unacceptable toxicity. All patients undergo surgical resection of the tumor on approximately day 21.

PROJECTED ACCRUAL: A total of 100 patients (25 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) of the breast

  * T0 disease
  * Newly diagnosed disease by minimally invasive biopsy (e.g., a vacuum-assisted large core tool [mammotome] or an equivalent method)
* Biopsy tissue available for molecular marker analysis
* Baseline mammography performed within the past 8 weeks
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, as defined by 1 of the following:

  * Age ≥ 60
  * Age ≥ 45 AND amenorrheic for > 1 year with uterus intact
  * Underwent bilateral oophorectomy
  * Follicle-stimulating hormone and estradiol levels in postmenopausal range

Performance status

* SWOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* SGOT and/or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 2.0 times ULN

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No history of deep vein thrombosis

Pulmonary

* No history of pulmonary embolism

Other

* Negative pregnancy test (if clinically indicated)
* No peripheral neuropathy > grade 1
* No underlying medical, psychiatric, or social condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 6 months since prior hormonal therapy, including any of the following:

  * Antiestrogens
  * Estrogen
  * Selective estrogen-receptor modulators
  * Progestins
  * Aromatase inhibitors

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for DCIS

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Molecular markers of the estrogen pathway as measured by immunohistochemistry at 3 weeks

SECONDARY OUTCOMES:
Mammographic breast density as measured by the Madena method at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California, United States